CLINICAL TRIAL: NCT01796899
Title: A Randomized, Single-center, Open-label, 5-way Crossover, Single-dose Bioavailability/Bioequivalence Comparison of Brivaracetam Oral Tablets (10 mg, 50 mg,75 mg, and 100 mg) and Brivaracetam Intravenous Bolus Injection (100 mg) in Healthy Volunteers
Brief Title: Comparison of Brivaracetam Oral Tablet (10 mg, 50 mg, 75 mg and 100 mg) and Brivaracetam Injection (100 mg) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: EP0007; 2012-001358-25 (EudraCT Number)
Record Dates: First submitted 2013-02-19; First posted 2013-02-22 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Brivaracetam
MeSH Terms: interventions — brivaracetam; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Brivaracetam 10 mg oral tablet (Other): Subjects check into the clinic the afternoon prior to the day of Brivaracetam (BRV) administration. The next day, a single dose of BRV 10 mg oral tablet will be administered in the morning. Following BRV administration, subjects will be observed for up to 48 hours. A Wash-Out Period of at least 7 days will separate the subsequent drug administrations.
  * Strength: 10 mg
  * Form: Oral tablet
  * Frequency: Once daily
  * Duration: 1 day
  Interventions: Other: Brivaracetam 10 mg oral tablet
- Brivaracetam 50 mg oral tablet (Other): Subjects check into the clinic the afternoon prior to the day of Brivaracetam (BRV) administration. The next day, a single dose of BRV 50 mg oral tablet will be administered in the morning. Following BRV administration, subjects will be observed for up to 48 hours. A Wash-Out Period of at least 7 days will separate the subsequent drug administrations.
  * Strength: 50 mg
  * Form: Oral tablet
  * Frequency: Once daily
  * Duration: 1 day
  Interventions: Other: Brivaracetam 50 mg oral tablet
- Brivaracetam 75 mg oral tablet (Other): Subjects check into the clinic the afternoon prior to the day of Brivaracetam (BRV) administration. The next day, a single dose of BRV 75 mg oral tablet will be administered in the morning. Following BRV administration, subjects will be observed for up to 48 hours. A Wash-Out Period of at least 7 days will separate the subsequent drug administrations.
  * Strength: 75 mg
  * Form: Oral tablet
  * Frequency: Once daily
  * Duration: 1 day
  Interventions: Other: Brivaracetam 75 mg oral tablet
- Brivaracetam 100 mg oral tablet (Other): Subjects check into the clinic the afternoon prior to the day of Brivaracetam (BRV) administration. The next day, a single dose of BRV 100 mg oral tablet will be administered in the morning. Following BRV administration, subjects will be observed for up to 48 hours. A Wash-Out Period of at least 7 days will separate the subsequent drug administrations.
  * Strength: 100 mg
  * Form: Oral tablet
  * Frequency: Once daily
  * Duration: 1 day
  Interventions: Other: Brivaracetam 100 mg oral tablet
- 10 mL of Brivaracetam intravenous bolus injection (10 mg/mL) (Other): Subjects check into the clinic the afternoon prior to the day of Brivaracetam (BRV) administration. The next day, a single dose of 10 mL of BRV intravenous bolus injection (10 mg/mL) will be administered in the morning. Following BRV administration, subjects will be observed for up to 48 hours. A Wash-Out Period of at least 7 days will separate the subsequent drug administrations.
  * Strength: 100 mg (10 mg/mL)
  * Form: Intravenous bolus injection
  * Frequency: Once daily
  * Duration: 1 day
  Interventions: Other: 10 mL of Brivaracetam intravenous bolus injection (10 mg/mL)

INTERVENTIONS:
Other: Brivaracetam 10 mg oral tablet
  Arms: Brivaracetam 10 mg oral tablet
Other: Brivaracetam 50 mg oral tablet
  Arms: Brivaracetam 50 mg oral tablet
Other: Brivaracetam 75 mg oral tablet
  Arms: Brivaracetam 75 mg oral tablet
Other: Brivaracetam 100 mg oral tablet
  Arms: Brivaracetam 100 mg oral tablet
Other: 10 mL of Brivaracetam intravenous bolus injection (10 mg/mL)
  Arms: 10 mL of Brivaracetam intravenous bolus injection (10 mg/mL)

SUMMARY:
To investigate the bioavailability/bioequivalence of Brivaracetam oral tablets (10 mg, 50 mg, 75 mg and 100 mg) and Brivaracetam intravenous injection (100 mg) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy male or female volunteer aged 18-55 years inclusive
* Subject has a Body Mass Index (BMI) of 18.0 - 30.0 kg/m^2 and a weight of at least 50 kg (males) or 45 kg (females)
* Subject has normal vital signs values, Electrocardiograms (ECGs) and clinical laboratory values
* Female subjects should have a negative pregnancy test or be of non-childbearing potential

Exclusion Criteria:

* Volunteer has participated or is participating in any other clinical studies of investigational drug or another Investigational Medicinal Product (IMP) within the last 3 months
* Volunteer is not healthy (eg, taking any drug treatments, excessive amount of alcohol, cigarettes or caffeine, having any medical or emotional/psychological problems, a drug/alcohol abuse, having abnormal safety parameters)
* Subject has an intolerance or allergy against the compound or related drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of Brivaracetam dose-normalized to the 50 mg reference treatment (Cmax) | Pharmacokinetic samples will be taken predose and 5 min, 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 6 h, 9 h, 12 h, 24 h, 36 h, and 48 h post dose
Area under the plasma concentration-time curve from zero to the time of the last measured concentration above the limit of quantification dose-normalized to the 50 mg reference treatment (AUC[0-t]) | Pharmacokinetic samples will be taken predose and 5 min, 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 6 h, 9 h, 12 h, 24 h, 36 h, and 48 h post dose
Area under the plasma concentration-time curve from zero to infinity dose-normalized to the 50 mg reference treatment (AUC) | Pharmacokinetic samples will be taken predose and 5 min, 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 6 h, 9 h, 12 h, 24 h, 36 h, and 48 h post dose

SECONDARY OUTCOMES:
Plasma half-life of Brivaracetam | Pharmacokinetic samples will be taken predose and 5 min, 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 6 h, 9 h, 12 h, 24 h, 36 h, and 48 h post dose
Time to reach the maximum plasma concentration of Brivaracetam (tmax) | Pharmacokinetic samples will be taken predose and 5 min, 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 6 h, 9 h, 12 h, 24 h, 36 h, and 48 h post dose
Apparent oral clearance of Brivaracetam (CL/F) | Pharmacokinetic samples will be taken predose and 5 min, 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 6 h, 9 h, 12 h, 24 h, 36 h, and 48 h post dose
Apparent volume of Brivaracetam distribution at the terminal elimination phase | Pharmacokinetic samples will be taken predose and 5 min, 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 6 h, 9 h, 12 h, 24 h, 36 h, and 48 h post dose

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 1, Zuidlaren, Netherlands